CLINICAL TRIAL: NCT03469960
Title: A Randomized Phase 3 Trial Comparing Continuation Nivolumab-Ipilimumab Doublet Immunotherapy Until Progression Versus Observation in Treatment-naive Patients With PDL1-positive Stage IV Non-Small Cell Lung Cancer (NSCLC) After Nivolumab-Ipilimumab Induction Treatment
Brief Title: Double Immune Checkpoint Inhibitors in PD-L1-positive Stage IV Non-small Lung CancEr
Acronym: DICIPLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1701; 2017-002540-33 (EudraCT Number)
Record Dates: First submitted 2018-02-16; First posted 2018-03-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
Keywords: IFCT; DICIPLE; NSCLC
MeSH Terms: interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : standard treatment (Active Comparator): 6 months of treatment by nivolumab + ipilimumab then nivolumab + ipilimumab then in case of progression platinum-based doublet recommended
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Arm B : experimental arm (Experimental): 6 months of treatment by nivolumab + ipilimumab then observation the in case of progression nivolumab + ipilimumab then in case of progression platinum-based doublet recommended
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 1 mg/kg every 6 weeks
Drug: Nivolumab — Nivolumab 3 mg/kg every 2 weeks

SUMMARY:
Non Small Cell lung cancer (NSCLC) remains the first cause of death by cancer in the World. For the patients presenting a NSCLC stage IV, the median of survival is about 15 months today. The chemotherapy with platinum is the standard treatment for these patients but immunotherapy showed these efficacy in 1st line for patients PD-L1 positive. On the other hand, the duration of treatment by immunotherapy is not clear. Indeed, prolonged responses and long survivals have been described in patients having interrupted the treatment. In the melanoma, a treatment of 6 months of ipilimumab demonstrated its efficacy. The objective of the study is to demonstrate that a treatment of 6 months followed by an observation (stop and go) is not less effective than a treatment given until progression or toxicity. This strategy would allow to decrease the accumulated toxicities, to improve the quality of life of the patients and to decrease the costs.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent:

   Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.

   Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
2. Histologically-proven NSCLC (squamous or non-squamous)
3. Stage IV (M1, including M1a pleural involvement) disease (8th classification TNM, UICC 2015)
4. ECOG PS < 1
5. Weight loss< 10% in previous 3 months
6. No prior systemic anticancer therapy (including EGFR or ALK inhibitors) given as primary therapy for advanced or metastatic disease.
7. Age≥ 18 years, <75 years
8. Life expectancy > 3 months
9. Measurable tumor disease by CT or MRI per RECIST 1.1 criteria
10. Available tumor samples for centralized PD-L1 immunohistochemistry analysis
11. PD-L1 tumor content ≥ 1% and < 50% tumor cells as assessed locally by the investigator center
12. Adequate biological functions:

    Creatinine Clearance ≥ 50 mL/min (Cockcroft or MDRD or CKD-epi); neutrophiles ≥ 1500/mm3 ; platelets ≥100 000/mm3 ; Hemoglobin ≥ 9g/dL ; hepatic enzymes < 3x ULN, total bilirubin ≤ 1,5 x ULN except for patients with proved, Gilbert syndrome (≤ 5 x ULN) or patients with hepatic metastases (≤ 3,0 mg/dL)
13. Women of childbearing potential (WOCBP) and sexually active should use an efficacious contraception method within the 28 days preceding the first dose and during the 6 months following the last dose of treatment. Women must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.

    For Male subjects who are sexually active with WOCBP, an efficacious contraception method should be used during the treatment and during the 7 months following the last dose.

    Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective.
14. Patient inclusion validated by a multidisciplinary meeting.

Exclusion Criteria:

1. Small cell lung cancer or tumors with mixt histology including a SCLC component
2. Known EGFR activating tumor mutation (deletion LREA in exon 19, L858R ou L861X mutations in exon 21, G719A/S mutation in exon 18) or HER exon 20 insertion (either tissue or plasma cfDNA mutation).
3. Known ALK or ROS1 gene rearrangement as assessed by immunohistochemistry, FISH or NGS sequencing
4. Previous or active cancer within the previous 5 years (except for treated carcinoma in situ of the cervix or basal cell skin cancer). Patients with a prostate adenocarcinoma history within the previous 5 years could be included in case of localized prostate cancer, with good prognostic factors according to d'Amico classification (≤ T2a and Score de Gleason ≤ 6 and PSA (ng/ml) ≤ 10), provided they were treated in a curative way (surgery or radiotherapy, without any chemotherapy)
5. Superior vena cava (SVC) syndrome persisting after SVC stenting
6. Thoracic radiotherapy needed at initiation of tumor treatment, except bone palliative radiotherapy on a painful or compressive metastasis, respecting 4 weeks delay between the end of radiotherapy and the beginning of induction immunotherapy treatment
7. Symptomatic untreated brain metastasis (without previous whole brain radiotherapy or stereotactic ablative brain radiotherapy or without surgical resection). At least 4 weeks delay between the end of radiotherapy and the beginning of induction immunotherapy treatment should be respected. Asymptomatic brain metastasis, not needing corticosteroids greater than 10 mg prednisone equivalent daily or mannitol infusions, with no evolution on brain MRI or CT-scan within the previous month are allowed.
8. History of previous primary immunodeficiency, organ transplantation needing an immunosuppressive treatment, any immunosuppressive drug within 28 days before randomization date, or history of severe toxicity (grade 3/4) by immune mechanism linked to another immunotherapy treatment.
9. Systemic treatment with corticosteroids with greater dose than 10 mg prednisone equivalent daily, within 14 days before initiation of the immunotherapy induction. Inhaled, nasal or topic corticosteroids are allowed.
10. History of active autoimmune disease including rheumatoid polyarthritis, Lupus, Wegener disease. Patients with type I diabetes, or hypothyroidism, or immune cutaneous disease (vitiligo, psoriasis, alopecia) not needing any immunosuppressive systemic treatment, are allowed to be included.
11. Active inflammatory intestinal disease (diverticulosis, Crohn disease, Hemorrhagic recto-colitis, coeliac disease) or any serious chronic intestinal disease with uncontrolled diarrhea
12. Active uncontrolled infection including tuberculosis, known acute viral hepatitis B and C according to serological tests. Patients with serological sequelae of cured viral hepatitis are allowed to be included.
13. HIV known infection
14. Living attenuated vaccine received within the 30 previous days
15. Previous treatment with anti-PD-1, anti-PD-L1 or Anti-CTLA4 antibody
16. Previous treatment with chemotherapy
17. General serious condition such as congestive uncontrolled cardiac failure, uncontrolled cardiac arrythmia, uncontrolled ischemic cardiac disease (unstable angina or history of myocardial infarction in the previous 6 months), history or stroke within the 6 previous months
18. Pre-existing lung interstitial disease as assessed by the diagnosis CT-scan.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS1) | 24 months after randomization of the last subject
  Time between the date of randomization and the first date of documented progression, as determined by BICR (Blinded Independent Central Review), or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS2) | 24 months after randomization of the last subject
  Time between the start date of the second line and the second date of documented progression, as determined by BICR, or death due to any cause, whichever occurs first.
Quality of life (QoL) | 24 months after randomization of the last subject
  Time until definitive deterioration (TUDD) from the randomization time in the experimental arm B.
Overall survival (OS) | 6, 12 and 18 months after randomization
Biological correlative exploratory studies (PD-L1) | 6 months
  PD-L1-stained % of tumor cells will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS
Biological correlative exploratory studies (PD-L1 H score) | 6 months
  PD-L1 H-score will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS
Biological correlative exploratory studies (CD3/CD8) | 6 months
  CD3/CD8 tumor infiltration will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS
Biological correlative exploratory studies (neutrophil) | 6 months
  neutrophil tumor infiltration will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS
Biological correlative exploratory studies (cytokines) | 6 months
  plasma concentration of different cytokines at baseline or at the randomization point, will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS
Biological correlative exploratory studies (chemokines) | 6 months
  plasma concentration of different chemokines at baseline or at the randomization point, will be associated to the rate of disease control patients at 6 months, PFS1, PFS2 and OS

CONTACTS AND LOCATIONS:
Locations (47):
- France (47):
  - Amiens - CHU, Amiens
  - Angers - CHU, Angers
  - Annecy - CH, Annecy
  - Argenteuil -CH, Argenteuil
  - Avignon - CH, Avignon
  - Bordeaux - Polyclinique Nord, Bordeaux
  - Boulogne - Ambroise Paré, Boulogne-Billancourt
  - Caen - CHU Côte de Nacre, Caen
  - Cahors - CH, Cahors
  - CH de Pontoise, Cergy-Pontoise
  - CH Chambery, Chambéry
  - CH de Chauny, Chauny
  - CH, Cholet
  - Clamart - Hôpital Percy, Clamart
  - Clermont Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Dijon - CAC, Dijon
  - CHRU Grenoble, Grenoble
  - La Roche Sur Yon - CH, La Roche-sur-Yon
  - Centre Hospitalier - Pneumologie, Le Mans
  - CHRU de Lille, Lille
  - CHU de Limoges, Limoges
  - CH Lyon Sud - Pneumologie, Lyon
  - Institut Paoli Calmette, Marseille
  - Marseille - Hôpital Européen, Marseille
  - Mont de Marsan - CH, Mont-de-Marsan
  - Mulhouse - CH, Mulhouse
  - Nantes - Centre René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Nîmes, Nîmes
  - Orléans - CH, Orléans
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - AP-HP Hôpital Bichat, Paris
  - GH Paris Saint-Joseph, Paris
  - Hôpital Saint Louis APHP, Paris
  - Paris - Institut Curie, Paris
  - Rouen - CHU, Rouen
  - Centre René Huguenin, Saint-Cloud
  - HIA Begin, Saint-Mandé
  - ICL Lucien Neuwirth, Saint-Priest-en-Jarez
  - Saint Quentin - CH, Saint-Quentin
  - Suresnes - Hopital Foch, Suresnes
  - Toulon - CHI, Toulon
  - CHU Toulouse, Toulouse
  - CHRU de Tours, Tours
  - Versailles - CH, Versailles
  - CH de Villefranche - Pneumologie, Villefranche

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data underlying the results reported in this article, as well as the study protocol and statistical analysis plan, will be made available after deidentification immediately following publication and for three years. Researchers who provide a methodologically sound proposal for any purpose may direct proposals to contact@ifct.fr. To gain access, data requestors will need to sign a data access agreement that requires approval by the French Cooperative Thoracic Intergroup.

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/151-ifct-1701